CLINICAL TRIAL: NCT01561040
Title: Eight Week Feasibility Study Enrolling Dry Eye Subjects Confirmed by Four of Seven Dianostic Markers Responding to Nutritional Therapy
Brief Title: Oral Nutrition Impact on Tear Film
Acronym: ONIT
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Eye and Vision Technologies and Research Institute (Network)
Collaborators: ZeaVision, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C-09-2011
Record Dates: First submitted 2011-10-25; First posted 2012-03-22 (Estimated); Last update posted 2012-03-26 (Estimated); Status verified 2012-03

CONDITIONS: Dry Eye Syndrome
Keywords: Dry Eye syndrome; tear film deficiency; Essential Fatty Acid nutritional supplements; Omega three supplements
MeSH Terms: conditions — Dry Eye Syndromes | interventions — Docosahexaenoic Acids

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Omega 3, Vitamins A, D3 and E (Experimental): Dry eye patients that have been screened with elevated osmolarity dispensed EZ Tears supplements containing Omega 3, Vitamins A, D3 and E to evaluate the change in dry eye conditions subjectively and objectively.
  Interventions: Dietary Supplement: Omega 3, Vitamins A, D3 and E

INTERVENTIONS:
Dietary Supplement: Omega 3, Vitamins A, D3 and E — omega 3 1480 mg vitamin A 1,000 IU vitamin D3 2,000 IU vitamin E 60 IU
  Other Names: EZ Tears

SUMMARY:
Dry eye disease (DED) is a common but often inadequately treated disease of the tears and surface of the eye. It can cause poor vision and chronic pain and is more frequent with increasing age. The 1995 Report of the National Eye Institute/Industry Workshop on Clinical Trials in Dry Eye defined dry eye as "a disorder of the tear film due to tear deficiency or excessive evaporation, which causes damage to the interpalpebral ocular surface and is associated with symptoms of ocular discomfort". The International Dry Eye Work Shop (DEWS) committee subsequently defined dry eye as "a multi-factorial disease of the tears and ocular surface that results in symptoms of discomfort, visual disturbance, and tear film instability with potential damage to the ocular surface. It is accompanied by increased osmolarity of the tear film and inflammation of the ocular surface." Typically, symptoms associated with dry eye disease include ocular burning, foreign body sensation (sand or grit), photophobia (light sensitivity), and other symptoms that result in overall long term discomfort in patients. The proposed eight week feasibility study if dry eye subjects confirmed elevated osmolarity and symptoms respond to nutritional therapy.

DETAILED DESCRIPTION:
Hyperosmolarity is a major cause of cell damage over time and can result in apoptosis of corneal and conjunctival cells. Determining if a patient has hyperosmolarity is critical allowing us to offer therapies to correct the problem. Reducing and regulating osmolarity is important in preventing potential long-term tissue compromise. Treatment leading to decreasing tear osmolarity can improve the patient's quality of life by stabilizing vision and, in many cases, simply allowing patients to return to normal activities.

Fatty Acids (EFA) have been shown to diminish inflammatory responses in many human inflammatory diseases, and interest in the use of omega-3 and omega-6 fatty acids for disease treatment has resulted in several small studies as well as the use (and over-the-counter availability) of EFA-containing nutritional supplements, including several specifically for the treatment of DED. Unfortunately, the effects of Omega 3 on dry eye disease have not been established to date. The purpose of this study is to better understand the role of Omega 3 plays in the regulating tear osmolarity in patients with established findings consistent with dry eye disease.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 79 at the time of informed consent.
* Must understand; be willing and able, and likely to fully comply with study procedures, visit schedule, and restrictions.
* A diagnosis of dry eye disease based on a global clinical assessment by the attending clinician, patient complaint of dry eye symptoms and osmolarity. There will be two osmolarity tiers; the lower tier is an open label design based on an average osmolarity between 316-326 mOsmo/L, and the other a group >=327 mOsmol/L. (Enrollment in the two tiers can either be simultaneous, or the second tier can be included after a responder analysis is done of tier 1).

Exclusion Criteria:

* Clinically significant eyelid deformity or eyelid movement disorder that is caused by conditions such as notch deformity, incomplete lid closure, entropion, ectropion, hordeola or chalazia.
* Previous ocular disease leaving sequelae or requiring current topical eye therapy other than for DED, including, but not limited to: active corneal or conjunctival infection of the eye and ocular surface scarring.
* Active ocular or nasal allergy.
* LASIK or PRK surgery that was performed within one year of Visit 1 or at any time during the study.
* Ophthalmologic drop use within 2 hours of any study visits.
* Pregnancy or lactation at any time during the study by history.
* Abnormality of nasolacrimal drainage (by history).
* Punctal cauterization or current punctal plug placement or within 30 days of punctual plug removal.
* Permissible Medications/Treatments- any commercially available OTC artificial tear.
* Prohibited Medications- Cyclosporine; any topical prescription medications (i.e., steroids, NSAIDs, etc); glaucoma medications; oral tetracyclines or topical macrolides; oral nutraceuticals (flax, fish, black currant seed oils, etc...) within 3 weeks of baseline.

Started or changed the dose of chronic systemic medication known to affect tear production including, but not limited to antihistamines, antidepressants, diuretics, corticosteroids or immunomodulators within 30 days of Visit 1.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2012-03; Primary Completion 2012-06 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Dry eye subjects ingesting omega three and the effect on seven diagnostic markers responding to omega 3 nutritional therapy. | two months
  This multi-centre study will screen patients with dry eye disease defined by objective diagnostic procedures to include TearLab Osmolarity, Tear Break Up Time (TBUT), Corneal Staining, Conjunctival Staining, phenol red thread test, Ocular Surface Disease Index and Meniscus height. Patients will also be assessed using subjective questionnaires to document the change of comfort and vision with the addition to their diet omega 3 supplements.

CONTACTS AND LOCATIONS:
Overall Officials: Sean Mulqueeny, OD, Principal Investigator; Robert L Davis, O.D., Study Director
Locations (4):
- United States (4):
  - Scot Morris, Conifer, Colorado
  - Davis EyeCare, Oak Lawn, Illinois
  - Koffler Vision Group, Lexington, Kentucky
  - Sean Mulqueeny OD, Creve Coeur, Missouri

REFERENCES:
- [Background] Png E, Samivelu GK, Yeo SH, Chew J, Chaurasia SS, Tong L. Hyperosmolarity-mediated mitochondrial dysfunction requires Transglutaminase-2 in human corneal epithelial cells. J Cell Physiol. 2011 Mar;226(3):693-9. doi: 10.1002/jcp.22389. PMID 20717931
- [Result] Sullivan BD, Whitmer D, Nichols KK, Tomlinson A, Foulks GN, Geerling G, Pepose JS, Kosheleff V, Porreco A, Lemp MA. An objective approach to dry eye disease severity. Invest Ophthalmol Vis Sci. 2010 Dec;51(12):6125-30. doi: 10.1167/iovs.10-5390. Epub 2010 Jul 14. PMID 20631232
- [Result] Chen Z, Tong L, Li Z, Yoon KC, Qi H, Farley W, Li DQ, Pflugfelder SC. Hyperosmolarity-induced cornification of human corneal epithelial cells is regulated by JNK MAPK. Invest Ophthalmol Vis Sci. 2008 Feb;49(2):539-49. doi: 10.1167/iovs.07-0569. PMID 18234997
- [Result] Suzuki M, Massingale ML, Ye F, Godbold J, Elfassy T, Vallabhajosyula M, Asbell PA. Tear osmolarity as a biomarker for dry eye disease severity. Invest Ophthalmol Vis Sci. 2010 Sep;51(9):4557-61. doi: 10.1167/iovs.09-4596. Epub 2010 Apr 14. PMID 20393114
- [Result] Versura P, Profazio V, Campos EC. Performance of tear osmolarity compared to previous diagnostic tests for dry eye diseases. Curr Eye Res. 2010 Jul;35(7):553-64. doi: 10.3109/02713683.2010.484557. PMID 20597641